CLINICAL TRIAL: NCT02524275
Title: Phase II Study of Docetaxel and Capecitabine in Advanced Squamous Cell Carcinoma of the Head and Neck
Brief Title: Docetaxel and Capecitabine With Recurrent or Metastatic Squamous Cell Carcinoma of the Head and Neck
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: low enrollment
Sponsor: University of Nebraska (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0762-14-FB; NCI-2015-00587 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2015-08-12; First posted 2015-08-14 (Estimated); Results first posted 2022-09-01 (Actual); Last update posted 2023-09-08 (Actual); Status verified 2023-08

CONDITIONS: Head and Neck Squamous Cell Carcinoma
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck | interventions — Capecitabine; Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (docetaxel, capecitabine) (Experimental): Patients receive docetaxel IV over 1 hour on day 1 and capecitabine PO BID on days 1-14. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Capecitabine; Drug: Docetaxel; Other: Quality-of-Life Assessment; Other: Questionnaire Administration

INTERVENTIONS:
Drug: Capecitabine — Given PO
  Other Names: Ro 09-1978/000; Xeloda
Drug: Docetaxel — Given IV
  Other Names: Docecad; RP56976; Taxotere; Taxotere Injection Concentrate
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This phase II trial studies the side effects and how well docetaxel and capecitabine work in treating patients with squamous cell (thin, flat cells) carcinoma of the head and neck that has come back or spread to other places in the body. Drugs used in chemotherapy, such as docetaxel and capecitabine, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate in a phase II study the efficacy (the radiographic assessment of disease status after 2 cycles of therapy) of a combination of docetaxel and capecitabine in subjects with advanced squamous cell carcinoma of the head and neck who are not candidates for surgery or radiation therapy.

II. To evaluate the safety and toxicities of docetaxel and capecitabine in subjects with advanced squamous cell carcinoma of the head and neck.

III. To descriptively examine the effects of the combination of docetaxel and capecitabine on the quality of life of subjects with advanced squamous cell carcinoma of the head and neck.

OUTLINE:

Patients receive docetaxel intravenously (IV) over 1 hour on day 1 and capecitabine orally (PO) twice daily (BID) on days 1-14. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up for 30 days and then periodically thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven squamous cell carcinoma of the head and neck with measurable disease that is either recurrent after attempted cure with surgery and/or radiation therapy or newly diagnosed disease with distant metastases or incurable at diagnosis
* Performance status: Karnofsky score >= 70 or Eastern Cooperative Oncology Group (ECOG) 0-2
* Age 19 years or older (age of consent in Nebraska); age 18 years or older (applicable to states where the age of majority is 18)
* No prior chemotherapy for metastatic squamous cell carcinoma of the head and neck; subjects who have received chemotherapy as part of a multi-modality curative approach for head and neck cancer will be eligible as long as they have not received either docetaxel or capecitabine (or fluorouracil [5-FU]) as part of that regimen
* White blood cell (WBC) count >= 3,500/mm^3
* Platelet count >= 100,000/mm^3
* Serum creatinine less than 1.5 times the upper limits of normal
* Serum aspartate aminotransferase (AST) and alanine aminotransferase (ALT) less than 1.5 times the upper limits of normal
* Serum alkaline phosphatase less than 2.5 times the upper limits of normal
* Serum total bilirubin is less than or equal to the upper limits of normal
* Prothrombin time (PT) or international normalized ratio (INR), and partial thromboplastin time (PTT) =< 1.5 x upper limit of normal unless subject is receiving anticoagulants; if the subject is on anticoagulation therapy, levels should be within therapeutic range
* Women of reproductive potential must be non-pregnant and non-nursing and must agree to employ an effective barrier method of birth control throughout the study and for up to 6 months following treatment
* Women of child-bearing potential must have a negative pregnancy test within 7 days of initiating study; (no childbearing potential is defined as age 55 years or older and no menses for two years or any age with surgical removal of the uterus and/or both ovaries)
* The subject must be aware of the neoplastic nature of his/her disease and willingly provide written, informed consent after being informed of the procedure to be followed, the experimental nature of the therapy, alternatives, potential benefits, side-effects, risks, and discomforts

Exclusion Criteria:

* Prior chemotherapy for metastatic squamous cell carcinoma of the head and neck; subjects who have received chemotherapy as part of a multi-modality curative approach for head and neck cancer will be eligible as long as they have not received either docetaxel or capecitabine (or 5-FU) as part of that regimen
* Allergy to either of the study medications or 5-fluorouracil
* Simultaneous participation in other therapeutic clinical trials will not be allowed
* If a subject is receiving allopurinol/cimetidine/antivirals they must be discontinued prior to starting this protocol
* Prior malignancy, except for adequately treated basal cell or squamous cell carcinoma of the skin, or thyroid cancer; carcinoma in situ of the cervix or breast; prostate cancer of Gleason grade 6 or less with stable prostate-specific antigen (PSA) levels (gonadotropin-releasing hormone [GnRH] analogs or androgen receptor blockers acceptable); or other cancers from which the subject has been disease-free for at least five years
* Uncontrolled intercurrent illnesses including, but not limited to symptomatic congestive heart failure, severe oxygen dependent chronic obstructive pulmonary disease, unstable angina or uncontrolled cardiac arrhythmia that could jeopardize the subject?s ability to receive the chemotherapy described in the protocol safely
* Pregnant and nursing women are excluded from this study
* Inability to co-operate with the study visit schedule and other requirements of the protocol
* Any other clinically significant medical disease or condition laboratory abnormality or psychiatric illness that, in the Investigator?s opinion, may interfere with protocol adherence or a subject?s ability to give informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2015-03-30 (Actual); Primary Completion 2021-10-28 (Actual); Study Completion 2021-10-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Apar Ganti, MD, Principal Investigator — University of Nebraska
Locations (3):
- United States (3):
  - Faith Regional Health Services Carson Cancer Center, Norfolk, Nebraska
  - Omaha Veterans Administration Medical Center, Omaha, Nebraska
  - University of Nebraska Medical Center, Omaha, Nebraska

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment (Docetaxel, Capecitabine)
Started | 14
Completed | 9
Not Completed | 5
Not completed — not evaluable, completed less than 2 courses of chemotherapy. | 5

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Docetaxel, Capecitabine)
Number analyzed (Participants) | 14
Age, Continuous [Mean (Full Range); unit: years] | 65.5 [47 to 80]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 14
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 13
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 14

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate of Complete or Partial Response
Description: The response rates of complete or partial response rate as defined by the Response Evaluation Criteria for Solid Tumors at 15 weeks of a chemotherapy regimen involving docetaxel and capecitabine as front line therapy at 95% confidence interval. Complete Response (CR): the disappearance of all target lesions Partial Response (PR): at least a 30% decrease in the sum of the longest diameter of target lesions, taking as reference the baseline sum longest diameter
Time Frame: At 15 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Docetaxel, Capecitabine)
Number analyzed (Participants) | 14
Participants | 1

2. Secondary Outcome: Progression-free Survival
Description: The Kaplan-Meier method will be used to estimate time to event distributions for progression-free survival. Progression-free survival will be defined as from the first date of therapy until the first notation of clinical progression, relapse or death from any cause.
Time Frame: First date of therapy until the first notation of clinical progression, relapse or death from any cause, assessed up to 5 years
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Treatment (Docetaxel, Capecitabine)
Number analyzed (Participants) | 14
days | 211 [63 to 327]

3. Secondary Outcome: Survival
Description: The Kaplan-Meier method will be used to estimate time to event distributions for survival. Survival will be defined as from the first date of therapy until the date of death from any cause.
Time Frame: First date of therapy until the date of death from any cause, assessed up to 5 years
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Treatment (Docetaxel, Capecitabine)
Number analyzed (Participants) | 14
days | 264.5 [147 to 516]

ADVERSE EVENTS:
Time Frame: Adverse Events will be collected from the time the subject starts the study drugs and ending 30 days following the final chemotherapy. Subjects with stable or responsive disease will continue on therapy until progression. For this study no subjects continued therapy beyond 12 months.
Arm/Group | Treatment (Docetaxel, Capecitabine)
All-Cause Mortality (participants affected / at risk) | 5/14
Serious Adverse Events (participants affected / at risk) | 10/14
Other Adverse Events (participants affected / at risk) | 13/14
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Docetaxel, Capecitabine) (N=14)
febrile nuetropenia (Blood and lymphatic system disorders) | 5 (5)
White blood cell decreased (Investigations) | 4 (4)
dysphagia (Gastrointestinal disorders) | 1 (1)
Gastrointestinal disorder, Other (Gastrointestinal disorders) | 1 (1) — Odynophagia
Mucositis, oral (Gastrointestinal disorders) | 2 (2)
Abdominal infection (Infections and infestations) | 1 (1)
hypocalcemia (Metabolism and nutrition disorders) | 1 (1)
vomiting (Gastrointestinal disorders) | 1 (1)
Neutrophil count decreased (Investigations) | 2 (2)
dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Urinary tract infection (Infections and infestations) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 2 (2)
hypoglycemia (Metabolism and nutrition disorders) | 1 (1)
Non-cardiac chest pain (General disorders) | 1 (1)
Respiratory, thoracic and mediastinal disorders, Other (Respiratory, thoracic and mediastinal disorders) | 1 (1) — COPD Exacerbation
lung infection (Infections and infestations) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Treatment (Docetaxel, Capecitabine) (N=14)
colitis (Gastrointestinal disorders) | 1/1 (1)
anemia (Blood and lymphatic system disorders) | 8 (12)
diarrhea (Gastrointestinal disorders) | 5 (6)
fatigue (General disorders) | 3 (5)
hypocalcemia (Metabolism and nutrition disorders) | 2 (4)
hypophosphatemia (Metabolism and nutrition disorders) | 1 (1)
lymphocyte count decreased (Blood and lymphatic system disorders) | 3 (5)
mucositis oral (Gastrointestinal disorders) | 6 (8)
nausea (Gastrointestinal disorders) | 4 (5)
neutrophil count decreased (Blood and lymphatic system disorders) | 2 (2)
thromboembolic event (Vascular disorders) | 1 (1)
white blood cell decreased (Blood and lymphatic system disorders) | 2 (2)
acute kidney injury (Renal and urinary disorders) | 1 (1)
alopecia (Skin and subcutaneous tissue disorders) | 1 (1)
anxiety (Psychiatric disorders) | 1 (1)
aspartate aminotransferase increased (Investigations) | 1 (1)
ataxia (Nervous system disorders) | 1 (1)
back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
blood bilirubin increased (Investigations) | 1 (1)
constipation (Gastrointestinal disorders) | 2 (2)
cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
creatinine increased (Investigations) | 2 (2)
dehydration (Metabolism and nutrition disorders) | 2 (3)
dizziness (Nervous system disorders) | 1 (2)
dry mouth (Gastrointestinal disorders) | 1 (1)
dysphagia (Gastrointestinal disorders) | 2 (2)
dyspnea (Respiratory, thoracic and mediastinal disorders) | 3 (3)
endocrine disorder - Other (Endocrine disorders) | 1 (1) — Right Thyroid Nodule
epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
erythroderma (Skin and subcutaneous tissue disorders) | 1 (1)
fall (Injury, poisoning and procedural complications) | 1 (1)
gastrointestinal disorder - Other (Gastrointestinal disorders) | 1 (1) — taste alterations
gastrointestinal disorder - Other (Gastrointestinal disorders) | 1 (1) — cholelithiasis
headache (Nervous system disorders) | 1 (1)
hypercalcemia (Metabolism and nutrition disorders) | 1 (1)
hyperglycemia (Metabolism and nutrition disorders) | 6 (8)
hypoalbuminemia (Metabolism and nutrition disorders) | 7 (9)
hypokalemia (Metabolism and nutrition disorders) | 4 (4)
hypomagnesemia (Metabolism and nutrition disorders) | 2 (2)
hyponatremia (Metabolism and nutrition disorders) | 1 (1)
hypotension (Vascular disorders) | 1 (1)
insomnia (Psychiatric disorders) | 1 (1)
investigations - Other (Investigations) | 1 (1) — hemoptysis
alkaline phosphatase increased (Investigations) | 1 (2)
metabolism and nutrition disorder - Other (Metabolism and nutrition disorders) | 1 (1) — hyperbilirubinemia
metabolism and nutrition disorder - Other (Metabolism and nutrition disorders) | 1 (1) — blood urea nitrogen (BUN) increased
musculoskeletal and connective tissue disorder - Other (Musculoskeletal and connective tissue disorders) | 1 (1) — Osteopenia
myalgia (Musculoskeletal and connective tissue disorders) | 1 (1)
nervous system disorder - Other (Nervous system disorders) | 1 (1) — leg cramps
non-cardiac chest pain (General disorders) | 2 (2)
oral pain (Gastrointestinal disorders) | 1 (1)
pain (General disorders) | 1 (1)
palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 3 (5)
palpitations (Cardiac disorders) | 1 (1)
peripheral sensory neuropathy (Nervous system disorders) | 1 (2)
platelet count decreased (Blood and lymphatic system disorders) | 2 (2)
pruritus (Skin and subcutaneous tissue disorders) | 1 (1)
rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1)
renal calculi (Renal and urinary disorders) | 1 (1)
respiratory, thoracic and mediastinal disorder - Other (Respiratory, thoracic and mediastinal disorders) | 1 (1) — viral infection - influenza B
skin and subcutaneous tissue disorder - Other (Skin and subcutaneous tissue disorders) | 1 (1) — desquamation over testicles
skin and subcutaneous tissue disorder - Other (Skin and subcutaneous tissue disorders) | 1 (1) — hand and foot syndrome
skin and subcutaneous tissue disorder - Other (Skin and subcutaneous tissue disorders) | 1 (1) — groin discoloration
skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 1 (1)
sore throat (Respiratory, thoracic and mediastinal disorders) | 1 (1)
stomach pain (Gastrointestinal disorders) | 1 (1)
tremor (Nervous system disorders) | 1 (1)
vomiting (Gastrointestinal disorders) | 3 (3)
wound dehiscence (Injury, poisoning and procedural complications) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-07-01): https://cdn.clinicaltrials.gov/large-docs/75/NCT02524275/Prot_SAP_000.pdf
  • Informed Consent Form (2021-01-21): https://cdn.clinicaltrials.gov/large-docs/75/NCT02524275/ICF_001.pdf